CLINICAL TRIAL: NCT07268300
Title: Breast Masses MRI Volumetry Compared to Post-operative Pathological Volume
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa kotb, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: BMRI-PATHVOL-TRIAL25
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Breast Masses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: Female patients aged between 18 and 65 years old. BIRADS classification IV, V, or VI with Operable breast cancer.

SUMMARY:
Breast cancer is one of the most common malignancies afflicting women worldwide 1.

Tumor size is important prognostic factor, its accurate measurement is essential for formulating surgery and chemotherapy plans. Additionally monitoring the change of tumor volume during treatment is an important for response evaluation criteria in solid tumors (RECIST) 1.

Typically, breast tumor size is reported from diameter measurements, using the unidimensional response evaluation criteria in solid tumors (RECIST) or the bidimensional WHO criteria. Both caliper techniques are widely employed methods for their simplicity 2. However, may be less sensitive than 3D volumetric measurement 3.

Breast cancers are less well circumscribed and more inhomogeneous on their border than benign lesions 2 and tumor necrosis correlated with tumor grade and aggressiveness is technically challenging while measuring tumor 1.

Measurements of tumor volume is more accurate than diameter and thus more sensitive to tumor size changes in response to treatment. 3D volume measurements more accurately capture the extent of irregularly shaped tumors, multifocality, and diffuse shrinkage of lesions during treatment 3.

Magnetic resonance imaging (MRI) is high resolution, inherent three-dimensionality and able to quantify tumor size 4,5. It is superior to mammography, sonography, and examination for revealing tumor extent in the breast and more accurately reflect the presence and size of residual disease after chemotherapy 3.

Previous studies investigated tumor size measured by the longest diameter on MRI agree with those on pathology 3.

Also 3D tumor volume correlation with those of other pathology has been investigated for was investigated in breast, prostate and pleural cancers 6-8 Our aim is to investigate CE-MRI tumor volume compared to pathology size.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged between 18 and 65 years old.
* BIRADS classification IV, V, or VI
* Operable breast cancer.
* 1st presentation.

Exclusion Criteria:

* Patients with contraindication for MRI imaging including heart pacemaker
* Patients with contrast media allergy.
* Prior history of breast cancer in the same breast with recurrence.
* Inflammatory carcinoma.
* Paget disease of the nipple

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: Female patients aged between 18 and 65 years old.BIRADS classification IV, V, or VI with Operable breast cancer.
Sampling Method: Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of MRI volumetry | baseline
  Accuracy of MRI volumetry of breast masses in estimating tumor volume